CLINICAL TRIAL: NCT05709925
Title: Effects of Instrument Assisted Soft Tissue Mobilization in Patients With Chronic Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/18
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomized Control Trial
Who Masked: Participant
Masking Description: Participants will be unaware of the type of the intervention they would be receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Group A will be receiving moist heat for 10 minutes followed by myofascial release through stripping technique to the lumbar region. After that post-treatment stretching would be performed. Total treatment plan would be of 30 minutes, comprising of total 9 sessions (3 weeks), 3 sessions on alternate days
  Interventions: Procedure: myofascial release
- Group B (Experimental): Group B will be receiving moist heat for 10 minutes followed by Instrument Assisted Soft Tissue Mobilization using long bar tool for 5-7 minutes with gentle horizontal stroking at an angle of 45 degrees. After that, post treatment stretching consisting of 2-3 sets of 10 repetitions of the targeted muscle group will be performed.Total treatment plan will be of 3 weeks comprising of total 9 sessions, 3 sessions on alternate days.
  Interventions: Procedure: Instrument Assisted Soft Tissue Mobilization

INTERVENTIONS:
Procedure: Instrument Assisted Soft Tissue Mobilization — The Graston Technique which is the Instrument Assisted Soft Tissue Mobilization is the use of a firm instrument to break tissue adhesions and mobilize scar tissue thus improving pain, range of motion and disability.
  Arms: Group B
Procedure: myofascial release — myofascial release through stripping technique to the lumbar region.
  Arms: Group A

SUMMARY:
This study is a Randomized Control Trial in which participants aged 18-50 years having diagnosed chronic mechanical low back pain will be recruited into two groups. Group A will be receiving myofascial release using stripping technique whereas, Group B will be receiving Instrument Assisted Soft Tissue Mobilization using long bar tool. Afterwards, post-treatment stretching would be performed in both the groups. Final assessment of pain, range of motion and disability will be done on last treatment session.

DETAILED DESCRIPTION:
Low Back Pain is a major cause of disability worldwide, affecting both genders equally at some point in their lives. 95% of low back pain is mechanical in origin which is the pain originating from spine, intervertebral discs and surrounding soft tissue structures. A total of 50 participants will be divided into two groups by coin toss method, based on the eligibility criteria. Baseline assessment of pain using NPRS, range of motion using Gravity-Based Inclinometer and disability using Oswestry Disability Index will be done on 1st session for both the groups. Group A will be receiving moist heat for 10 minutes followed by myofascial release and post-treatment stretching. Whereas, on the other hand, Group B will be receiving moist heat for 10 minutes followed by Instrument Assisted Soft Tissue Mobilization using Graston G6 long bar tool for 5-7 minutes with gentle horizontal stroking at an angle of 45 degrees over lumbar area followed by post-treatment stretching. Total treatment plan will be of 3 weeks, consisting of total 9 sessions, 3 sessions on alternate days. Final assessment will be done for pain, range of motion and disability on last session at 3rd week. Gentle icing would be recommended in case of itching and bruising over the treated area.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-50 years with diagnosed chronic mechanical low back pain.
* Males and females both.
* Participants having symptoms of duration more than 3 months.
* Numeric Pain Rating Scale (NPRS) score of 5 or more.

Exclusion Criteria:

* Patient with a history of recent spinal surgery and related trauma.
* Participants with a history of pregnancy.
* Participants with a history of infection, tumor and spinal fracture.
* Participants with diagnosed Psychiatric Disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar range of motion | 3 weeks
  Range of motion is the ability of a joint to go through its complete spectrum of movement and it will be measured using gravity-based inclinometer.

SECONDARY OUTCOMES:
Pain Intensity | 3 weeks
  Pain will be measured using Numeric Pain Rating Scale which is an eleven point scale scored from 0 indicating no pain and 10 indicating worst pain.
Lumbar Disability | 3 weeks
  Lumbar disability will be measured using Oswestry Disability Index which is a valid and reliable tool consisting of 10 items from which patient gets to choose according to their level of function.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan

REFERENCES:
- [Derived] Gul S, Bashir S, Kayani NM, Sabir Z, Qurat-Ul-Ain H. Effects of instrument assisted soft tissue mobilisation in patients with chronic mechanical low back pain----A randomized control trial. J Pak Med Assoc. 2025 Feb;75(2):181-185. doi: 10.47391/JPMA.11511. PMID 39948773